CLINICAL TRIAL: NCT04486599
Title: Feasibility of Electromagnetic Navigation During Ultrasound Guided Foam Sclerotherapy for the Treatment of Venous Malformations.
Brief Title: Electromagnetic Navigation During Ultrasound Guided Foam Sclerotherapy for Venous Malformations
Acronym: SCLERONAV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/19/0516
Record Dates: First submitted 2020-07-09; First posted 2020-07-24 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Venous Malformation
Keywords: Foam Sclerotherapy; Ultrasound; Electromagnetic Navigation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electromagnetic Navigation (Experimental): The patient have to low Flow Vascular Abnormality diagnosed by Duplex Ultrasound and MRI. Decision of Ultrasound Guided Percutaneous Foam Sclerotherapy taken in multidisciplinary staff meeting
  Interventions: Device: Electromagnetic Navigation

INTERVENTIONS:
Device: Electromagnetic Navigation — The echo-guided sclerotherapy procedure, assisted by electromagnetic navigation, will be carried out in a clean room during the day hospitalisation and followed by a control Echo-Doppler carried out 2 hours after the procedure.

SUMMARY:
The aim of this study is to evaluate the feasibility of assisted electromagnetic navigation in percutaneous echo-guided sclerotherapy of slow-flow vascular malformations. Feasibility will be defined in terms of the percentage of patients for whom the procedure is successful.

DETAILED DESCRIPTION:
Primary interventional treatment of low flow vascular anomalies includes ultrasound guided foam sclerotherapy. Each procedure involves a percutaneous needle insertion. However, procedures remain complicated to obtain the right trajectory in order to inject the foam at the center of the abnormality. Electromagnetic navigation system tracks the operator's needle, meaning the position and progression of the needle is visualized in 3D real time on the ultrasound probe interface.

The present trial evaluate the feasibility of the electromagnetic navigation system during the needle insertion and the improvement of needle placement accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Low Flow Vascular Abnormality diagnosed by Duplex Ultrasound and MRI
* Decision of Ultrasound Guided Percutaneous Foam Sclerotherapy taken in multidisciplinary staff meeting

Exclusion Criteria:

* patients with pacemakers or internal defibrillator
* patients with ferromagnetic implanted material
* patients who are wards of court or under guardianship
* patients deprived of freedom by judicial or administrative decision
* patients under legal protection
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients for whom the procedure is successful | day 1
  Success of procedure a.e. obtention of venous flow at the extremity of the needle permitting the realization of the foam sclerotherapy treatment.

SECONDARY OUTCOMES:
Estimate the number of punctures required to achieve catheterization of the malformation. | day 1
  Number of percutaneous punctures needed to obtain vascular backflow.
Estimate the time to complete catheterization of the malformation | day 1
  Duration of the procedure.
Estimate the undesirable effects associated with assisted electromagnetic navigation. | day 1
  Adverse effects of Electro-Magnetic Navigation.

CONTACTS AND LOCATIONS:
Overall Officials: Wassim Mokaddem, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital, Toulouse, Occitanie, France